CLINICAL TRIAL: NCT05363202
Title: A Randomized, Assessor-blind, Placebo Controlled, Multicenter, Clinical Endpoint Bioequivalence Study to Compare the Efficacy and Safety of Generic Fluticasone Propionate Inhalation Aerosol USP 44 mcg (Glenmark Pharmaceuticals Ltd) to Flovent HFA (Fluticasone Propionate Inhalation Aerosol) 44 mcg (GSK Group of Companies) in Treatment of Patients With Bronchial Asthma.
Brief Title: To Study Generic Fluticasone Propionate Inhalation Aerosol for the Treatment of Bronchial Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLK 2101
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Fluticasone propionate inhalation aerosol USP 44 mcg (Glenmark Pharmaceuticals Ltd.) (Experimental)
  Interventions: Drug: Fluticasone propionate Inhalation Aerosol 44 mcg
- FLOVENT HFA (Active Comparator)
  Interventions: Drug: FLOVENT HFA 44 mcg
- Placebo of Fluticasone propionate inhalation aerosol 44 mcg (Placebo Comparator)
  Interventions: Drug: Matching Placebo inhaler

INTERVENTIONS:
Drug: Fluticasone propionate Inhalation Aerosol 44 mcg — Dosage Form: Metered dose Inhalation Aerosol Dosage Frequency 44 mcg (two inhalations; twice daily (i.e. morning & evening approximately. 12 h apart, Mode of Administration: Oral inhalation
  Arms: Fluticasone propionate inhalation aerosol USP 44 mcg (Glenmark Pharmaceuticals Ltd.)
Drug: FLOVENT HFA 44 mcg — Dosage Form: Metered dose Inhalation Aerosol Dosage Frequency 44 mcg (two inhalations; twice daily (i.e. morning & evening approximately. 12 h apart, Mode of Administration: Oral inhalation
  Arms: FLOVENT HFA
Drug: Matching Placebo inhaler — Dosage Form: Metered dose Inhalation Aerosol Dosage Frequency 44 mcg (two inhalations; twice daily (i.e. morning & evening approximately. 12 h apart, Mode of Administration: Oral inhalation
  Arms: Placebo of Fluticasone propionate inhalation aerosol 44 mcg

SUMMARY:
This is a randomized, assessor-blind, placebo controlled, multicenter, clinical endpoint bioequivalence study to compare the efficacy and safety of generic fluticasone propionate inhalation aerosol USP 44 mcg (Glenmark Pharmaceuticals Ltd) to Flovent HFA (fluticasone propionate inhalation aerosol) 44 mcg (GSK group of companies) in treatment of patients with bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects aged between 18 to 65 years of age (both ages inclusive)
2. Diagnosis of asthma for at least 12 months prior to screening
3. Pre-bronchodilator FEV1 of more than or equal to 45 % and less than or equal to 85 %.
4. Subjects should be stable on their chronic asthma treatment regimen for at least 4 weeks prior to screening
5. Currently non-smoking;
6. More than or equal to 15 % reversibility of FEV1 within 30 min following 360 mcg of Albuterol/salbutamol inhalation (pMDI) at screening
7. Ability to discontinue their asthma controller medication safely
8. Ability to replace short-acting β agonists (SABAs) ongoing at screening with Albuterol/salbutamol inhaler.
9. Women of childbearing potential must be willing to consistently use an appropriate method of contraception.
10. Willingness to give their written informed consent to participate in the study.
11. Is willing to comply with all aspects of the protocol.
12. Ability to follow training given for study related procedures and assessments in the opinion of the Investigator.

Exclusion Criteria:

1. Patients with life-threatening asthma,
2. Significant respiratory disease other than asthma
3. Evidence or history of clinically significant medical, surgical or psychiatric disease or laboratory abnormalities.
4. Known hypersensitivity to any sympathomimetic drug.
5. Subjects receiving β2-blockers, anti-arrhythmics, anti-depressants, and/or monoamine oxidase inhibitors within 4 weeks prior to the screening.
6. Viral or bacterial, upper or lower respiratory tract infection, or sinus, or middle ear infection within 4 weeks prior to the screening visit
7. Subjects who required biologic agents for asthma systemic or oral corticosteroids (for any reason), within the past 6 months prior to screening
8. Evidence or history of oral candidiasis, active tuberculosis, hypercorticism, adrenal suppression, or eye problems.
9. Female subjects who are pregnant or breast-feeding or planning to be pregnant.
10. Currently enrolled in another clinical study or used any investigational product (study drug), study drug, or device within 30 days or 5 elimination half-lives, whichever is longer, preceding informed consent.
11. Consumes excessive amounts of alcohol, abuses drugs, or has any condition that would compromise compliance with this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
- Change from baseline in FEV1 measured in the morning prior to dosing of inhaled medications on the last day of 4-week treatment period | From Baseline to last day of 4-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Ameet Daftary, Study Director — Glenmark Pharmaceuticals Ltd
Locations (11):
- India (11):
  - Investigational Site 9, Ahmedabad, Gujarat
  - Investigational Site 2, Aurangabad, Maharashtra
  - Investigational Site 6, Nagpur, Maharashtra
  - Investigational Site 16, Nashik, Maharashtra
  - Investigational Site 11, Nashik, Maharashtra
  - Investigational Site 10, Nashik, Maharashtra
  - Investigational Site 3, Pune, Maharashtra
  - Investigational Site 1, Pune, Maharashtra
  - Investigational Site 4, Jaipur, Rajasthan
  - Investigational Site 13, Hyderabad, Telangana
  - Investigational Site 5, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No